CLINICAL TRIAL: NCT01080651
Title: Clinical Trials to Evaluate the Influence of CYP2C19 Genotype and Drug-drug Interactions on the Pharmacokinetics of Voriconazole in Healthy Korean Male Volunteers (Part B)
Brief Title: Influence of Drug-drug Interactions on the Pharmacokinetics (PK) of Voriconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: In-Jin Jang, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: SNUCPT09_Vori2C19_B
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Invasive Aspergillosis
MeSH Terms: interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CYP2C19 extensive metabolizer (Active Comparator)
  Interventions: Drug: Voriconazole
- CYP2C19 poor metabolizer (Active Comparator)
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — Day1: voriconazole 200 mg x 2, oral administration, Day2-7: rifampin 600 mg, once a day oral administration, Day8: voriconazole 200 mg x 2 + rifampin 600 mg, oral co-administration

SUMMARY:
To evaluate the drug-drug interaction between rifampicin and voriconazole according to CYP2C19 genotype quantitatively following a single oral administration of 200 mg voriconazole

ELIGIBILITY:
Inclusion Criteria:

* 1.Healthy male subjects aged 20 - 50 years.
* 2.A body mass index (BMI) in the range 17-28 kg/m2.
* 3.Sufficient ability to understand the nature of the study and any hazards of participating in it. Provide written informed consent after being fully informed about the study procedures.

Exclusion Criteria:

* 1.Presence or history of severe adverse reaction to any drug or a history of severe allergic disease.
* 2.Clinically relevant abnormal medical history that could interfere with the objectives of the study.
* 3.Presence or history of eye disease or eye field defect.
* 4.A subject with history of gastrointestinal disease or surgery (except simple appendectomy or repair of hernia), which can influence the absorption of the study drug.
* 5.A subject whose liver function test (AST, ALT, GGT, ALP, LDH) result is over 1.25 times of upper limit of normal range.
* 6.A subject whose SBP is over 140 mmHg or below 90 mmHg and DBP is over 100 mmHg or below 50 mmHg.
* 7.Presence or history of drug abuse.
* 8.Participation in other clinical trial within 2 months.
* 9.Use of a prescription medicine, herbal medicine within 2 weeks or over-the-counter medication within 1 week before first dose.
* 10.Blood donation during 2 months or apheresis during 1 month before the study.
* 11.Presence or history of alcohol abuse.
* 12.Smoking of more than 10 cigarettes/day.
* 13.Use of grapefruit juice, xanthine containing beverage, alcohol or smoking during restriction period.
* 14.Subject judged not eligible for study participation by investigator.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of voriconazole | pre-dose, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h post-dose
  Sample for concentration measurement conducted before and after rifampicin treatment as same manner

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, M.D., Ph.D., Principal Investigator — Professor
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea